CLINICAL TRIAL: NCT00527163
Title: Role of Nitric Oxide Scavenging by Plasma Hemoglobin and Identification of Hemolysis-Associated Pulmonary Hypertension in Malaria
Brief Title: Role of Nitric Oxide in Malaria
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907217; 07-H-N217
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2015-03-30

CONDITIONS: Malaria; Pulmonary Hypertension
Keywords: Echocardiogram; Endothelial Dysfunction; Malaria; Mali; Screening
MeSH Terms: conditions — Malaria; Hypertension, Pulmonary

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study, conducted by NIH, the University of Bamako in Mali, Africa, and Tulane University will examine the relationships between hemolysis (breakdown of red blood cells), nitric oxide (a gas important in regulating blood vessel dilation and blood flow) and pulmonary hypertension in patients with malaria. Malaria is among the leading causes of death in many of the world s poorest countries. It is caused by a parasite that is transmitted to humans by mosquitoes.

Malian children ages 1-5 years are eligible for participation in this study. They include children with asymptomatic infection, uncomplicated disease, and severe disease. Uninfected controls are also included.

Upon enrollment, participants have a medical history and physical examination, echocardiogram (ultrasound test of heart function) and blood tests. In addition, all participants (infected children and controls) have repeat evaluations when healthy, approximately 7 to10 days following successful therapy.

DETAILED DESCRIPTION:
Malaria is among the leading infectious causes of death in many of the world s poorest countries. This parasitic mosquito-borne illness produces massive hemolysis in many infected human hosts. While much is known about parasite replication and cytoadherence, very little is known about the impact of hemolysis per se on vascular tone and endothelial function. Crossing a number of medical disciplines beyond the scope of malaria, intriguing new research on inherited hemolytic disorders such as sickle cell disease (SCD) provides clues to pathogenic mechanisms that may be relevant to malaria. Dr. Gladwin (NHLBI) and colleagues have characterized a mechanism of disease, hemolysis-associated endothelial dysfunction, in which red blood cell hemoglobin spills into plasma and reacts with and oxidatively destroys nitric oxide (NO). Additionally, erythrocyte arginase I is released into plasma and catabolizes arginine, the substrate for endothelial NO synthesis. As a result, the profound reduction in NO bioavailability produces vasomotor instability, oxidant stress, inflammation, endothelial adhesion molecule expression, activation of tissue factor, and platelet aggregation. Consistent with shared mechanisms, these same pathways are found to be activated during malarial infection. Chronic hemolysis in hemoglobinopathies also leads to a disease syndrome, hemolysis associated pulmonary hypertension, which develops in all chronic hereditary and acquired hemolytic conditions and is associated with excessive morbidity and mortality. Despite the recent appreciation of these mechanisms, not one study can be found in the literature evaluating pulmonary hypertension in human malaria.

This protocol therefore aims to evaluate mechanisms governing interrelationships among malaria, intravascular hemolysis, NO bioavailability, endothelial function, pulmonary hypertension, and evolutionarily selected host polymorphisms that regulate the host response to hemolysis. We will correlate our clinical observations in the field with laboratory assays of hemolysis and nitric oxide bioavailability related to scavenging by cell-free hemoglobin and arginine catabolism. Using a candidate gene approach, we will identify and selectively characterize polymorphisms in genes important for endothelial function, vascular inflammation and disease phenotype. Finally, the characterization of this mechanism in malaria may catalyze the development of novel therapies targeting this pathway, such as sodium nitrite, inhaled nitric oxide gas, and/or recombinant haptoglobin infusions.

This international collaboration between scientists at the NIH, University of Bamako, and Tulane University will provide an exclusive opportunity for the rapid transfer of appropriate technology and expertise relevant to the provision of the highest quality care to malaria patients in Mali and the world.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Malian children ages 1-5 years are eligible for participation in this study. We require a parent or legally authorized guardian to be present at enrollment to provide consent. Given the eligibility ages for children, incipient maturity and intelligence do not permit direct participant assent.

INCLUSION CRITERIA:

Inclusion criteria for Healthy Uninfected controls:

* Malian children ages 1-5 years, regardless of gender or ethnicity.
* A peripheral blood smear negative for the presence of Plasmodium falciparum.
* Temperature less than or equal to 37.5 degrees Celsius.
* The child s parent or guardian must be present for consent and enrollment.

Inclusion criteria for Asymptomatic Parasitemia controls:

* Malian children ages 1-5 years, regardless of gender or ethnicity.
* Plasmodium falciparum microscopically visualized on blood smear, with asexual parasite density greater than or equal to 2,000/microL of blood and less than 500,000/microL of blood.
* Temperature less than or equal to 37.5 degrees Celsius.
* The child s parent or guardian must be present for consent and enrollment.

Inclusion criteria for Uncomplicated Malaria cases:

* Malian children ages 1-5 years, regardless of gender or ethnicity.
* Plasmodium falciparum microscopically visualized on blood smear, with asexual parasite density greater than or equal to 2,000/microL of blood and less than 500,000/microL of blood.
* Signs and symptoms of malaria (e.g. headache, body aches, malaise).
* Temperature 37.6 - 39.9 degrees Celsius, OR history of fever.
* The child s parent or guardian must be present for consent and enrollment.

Inclusion criteria for Severe Malarial Anemia cases:

* Malian children ages 1-5 years, regardless of gender or ethnicity.
* Plasmodium falciparum microscopically visualized on blood smear, with asexual parasite density greater than or equal to 2,000/microL of blood and less than 500,000/microL of blood.
* Hemoglobin less than 5 g/dL, or hemoglobin 5.0-6.9 g/dL if accompanied by respiratory distress.
* The child s parent or guardian must be present for consent and enrollment.

EXCLUSION CRITERIA:

Exclusion criteria for Healthy Uninfected controls:

* Signs or symptoms consistent with malaria (e.g. headache, body aches, malaise).
* Temperature greater than 37.5 degrees Celsius, OR history of fever.
* History of anti-malarial medication use within 2 weeks prior to enrollment.
* Transfusion of any blood products within 2 weeks prior to enrollment.
* Signs or symptoms of active infectious disease, whether bacterial, viral, or parasitic in nature.
* Co-existing severe or chronic medical conditions (e.g. bacteremia, meningitis, kwashiorkor, renal failure, recent trauma, etc.).

Exclusion criteria for Asymptomatic Parasitemia controls:

* Signs or symptoms consistent with malaria (e.g. headache, body aches, malaise).
* Temperature greater than 37.5 degrees Celsius, OR history of fever.
* History of anti-malarial medication use within 2 weeks prior to enrollment.
* Transfusion of any blood products within 2 weeks prior to enrollment.
* Signs or symptoms of active infectious disease, whether bacterial, viral, or parasitic in nature.
* Co-existing severe or chronic medical conditions (e.g. bacteremia, meningitis, kwashiorkor, renal failure, recent trauma, etc.).

Exclusion criteria for Uncomplicated Malaria cases:

* Any criteria of severe malaria, including:

  * CEREBRAL MALARIA Coma (Blantyre coma score less than or equal to or convulsions [witnessed by investigator]).
  * SEVERE ANEMIA (hemoglobin less than 5 g/dL).
  * RESPIRATORY DISTRESS (respiratory rate greater than 40 with 2 of the following: nasal flaring, intercostal indrawing, subcostal recession and grunting).
  * HYPOGLYCEMIA (blood glucose less than 40 mg/dL).
  * RENAL FAILURE (no urine output for 24 hours).
  * JAUNDICE/ICTERUS.
  * SEVERE PROSTRATION (if greater than 7 months old, inability to sit and drink).
  * HYPERPARASITEMIA (asexual parasite density greater than or equal to 500,000/microL of blood).
  * SHOCK (systolic blood pressure less than 50 mmHg, rapid pulse, cool extremities).
  * REPETITIVE VOMITING with cessation of eating and drinking.
  * HYPERPYREXIA (temperature greater than or equal to 40 degrees Celsius).
* Etiologies of febrile illness (e.g. respiratory tract infection, cellulitis) on clinical examination not attributable to malaria.
* Co-existing severe or chronic medical conditions (e.g. bacteremia, meningitis, kwashiorkor, renal failure, recent trauma, etc.) unrelated to P. falciparum infection.
* Transfusion of any blood products within 2 weeks prior to enrollment.

Exclusion criteria for Severe Malarial Anemia cases:

* Evidence of CEREBRAL MALARIA.

  * Coma (Blantyre coma score less than or equal to 2), or
  * Convulsions (witnessed by investigator).
* Evidence of HYPOGLYCEMIA.

  --Blood glucose less than 40 mg/dL.
* Evidence of HYPERPARASITEMIA.

  --Asexual parasite density greater than or equal to 500,000/microL of blood.
* Evidence of SHOCK.

  --Systolic blood pressure less than 50 mmHg with signs of hypoperfusion and circulatory collapse (e.g. rapid pulse, cool extremities).
* Etiologies of febrile illness (e.g. respiratory tract infection, cellulitis) on clinical examination that are not attributable to malaria.
* Co-existing severe or chronic medical conditions (e.g. bacteremia, meningitis, kwashiorkor, renal failure, recent trauma, etc.) unrelated to P. falciparum infection.
* Transfusion of any blood products within 2 weeks prior to enrollment.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2007-09-04; Study Completion 2015-03-30

CONTACTS AND LOCATIONS:
Overall Officials: Henry Masur, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- Hospital Gabriel Toure, Bamako, Mali

REFERENCES:
- [Background] Rother RP, Bell L, Hillmen P, Gladwin MT. The clinical sequelae of intravascular hemolysis and extracellular plasma hemoglobin: a novel mechanism of human disease. JAMA. 2005 Apr 6;293(13):1653-62. doi: 10.1001/jama.293.13.1653. PMID 15811985
- [Background] Kato GJ, Martyr S, Blackwelder WC, Nichols JS, Coles WA, Hunter LA, Brennan ML, Hazen SL, Gladwin MT. Levels of soluble endothelium-derived adhesion molecules in patients with sickle cell disease are associated with pulmonary hypertension, organ dysfunction, and mortality. Br J Haematol. 2005 Sep;130(6):943-53. doi: 10.1111/j.1365-2141.2005.05701.x. PMID 16156864
- [Background] Gladwin MT, Sachdev V, Jison ML, Shizukuda Y, Plehn JF, Minter K, Brown B, Coles WA, Nichols JS, Ernst I, Hunter LA, Blackwelder WC, Schechter AN, Rodgers GP, Castro O, Ognibene FP. Pulmonary hypertension as a risk factor for death in patients with sickle cell disease. N Engl J Med. 2004 Feb 26;350(9):886-95. doi: 10.1056/NEJMoa035477. PMID 14985486